CLINICAL TRIAL: NCT01205906
Title: Comparison of the Efficacy of an Internet-based Self-help Training and a Well-established Outpatient Group Therapy for the Treatment of Chronic Tinnitus: A Randomized Controlled Trial
Brief Title: Comparison of an Internet-based Guided Self-help and a Group Therapy for Chronic Tinnitus
Acronym: MINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Maria Kleinstäuber, Dr., Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MINT-100510
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2014-04

CONDITIONS: Tinnitus
Keywords: Tinnitus; Internet Training; Cognitive-Behavior Therapy; CBT
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Internet-based guided self-help (Experimental): This self-help training is exclusively provided via Internet over a period of 10 weeks. The treatment is based on the cognitive-behavioral approach and consists of 18 modules with helpful strategies to cope with tinnitus (e.g., applied relaxation, positive imagery, attention shift exercises, cognitive restructuring, sleep management, concentration management,). All modules include an information text, detailed practice instructions, worksheets and homework assignments. At the end of each treatment week, there is an e-mail contact between the participants and their therapist. The participants report on their work with the modules and if they had encountered any problems. The therapist provides feedback, support and recommendations on how to proceed.
  Interventions: Behavioral: Internet-based guided self-help for tinnitus
- Cognitive-behavior group therapy (Experimental): This well-established, cognitive-behavior group therapy was developed by Hiller and Haerkötter (2005) and consists of 10 weekly group sessions of 90 minutes. The strictly manualized program includes the following components focusing on the special needs of chronic tinnitus patients: Education, relaxation techniques, cognitive restructuring, the role of attentional processes for tinnitus perception, analysis of avoidance behaviors, tinnitus and the health care system as well as relapse prevention. For each session participants receive written materials, exercises and homework assignments to enhance understanding and to transfer the new information into the daily routine.
  Interventions: Behavioral: Cognitive-behavior group therapy for tinnitus
- Discussion forum group (Active Comparator): To the participants of the control group the group therapy or the internet-based self-help after waiting time of 10 weeks is offered. During the waiting period participants receive access to a tinnitus online discussion forum.
  Interventions: Other: Internet discussion forum

INTERVENTIONS:
Behavioral: Internet-based guided self-help for tinnitus — Internet-based self-help for tinnitus: provided via Internet, duration of 10 weeks
  Arms: Internet-based guided self-help
Behavioral: Cognitive-behavior group therapy for tinnitus — Cognitive-behavior group therapy for tinnitus: weekly group sessions of 90 minutes, duration of 10 weeks
  Arms: Cognitive-behavior group therapy
Other: Internet discussion forum — Tinnitus-specific internet discussion forum over 10 weeks (no therapeutic intervention)
  Arms: Discussion forum group

SUMMARY:
The aim of this study is to compare the efficacy of an internet-based guided self-help training for chronic tinnitus with a well-established outpatient group therapy and a discussion forum group.

DETAILED DESCRIPTION:
Chronic tinnitus can result in significant psychological suffering and reduce quality of life. Cognitive behavioral therapy (CBT) has been shown to be effective in decreasing the impairment caused by tinnitus. One recent way delivering CBT is an internet-based self-help intervention. Internet interventions for patients with chronic tinnitus, developed by Swedish scientists, showed promising results (Andersson et al., 2002; Kaldo et al., 2007; Kaldo et al., 2008). The main purpose of this study is to compare the efficacy of this internet-based self-help training for chronic tinnitus with a traditional well-established CBT group treatment and with a discussion forum group in a randomized controlled trial. Secondary goals are a process evaluation of both treatments, the identification of predictors of treatment success, an estimation of the cost-effectiveness of each treatment and the validation of the Tinnitus Cognitions Questionnaire (T-Cog; Hiller & Haerkötter, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Chronic tinnitus for at least 6 months
* Medical examination of tinnitus by an ear, nose and throat physician (ENT)
* Scoring 18 or above on the Tinnitus Handicap Inventory (THI) or scoring 12 or above in the Mini-Tinnitus Questionnaire (Mini-TQ)
* Not currently receiving psychological treatment for tinnitus
* Being able to access the Internet and print instructions
* Sufficient knowledge of the German language to read and follow the internet-based self-help training
* Being able to attend weekly group sessions in the Outpatient Department of the Psychological Institute of the University of Mainz, Germany
* Sufficient time and motivation to work on the treatment programs

Exclusion Criteria:

* Tinnitus caused by any other general medical condition or otologic disease (e.g., active Meniere's Disease)
* Clinical diagnosis of any severe mental disorder (especially a severe depressive disorder, suicidality, acute psychosis)
* Clinical diagnosis of Dementia or another severe organic cerebral disorder
* Clinical diagnosis of substance-related addiction/abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI; Newman, Jacobson, & Spitzer, 1996; German version: Kleinjung et al., 2007) | 18 months
  The measure assesses tinnitus-related disability and handicap.
MINI-Tinnitus Questionnaire (Mini-TQ; Hiller & Goebel, 2004) | 18 months
  The measure is a short version of the Tinnitus Questionnaire (TQ, Goebel & Hiller, 1998), to assess tinnitus-related psychological distress

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS-D; Zigmond & Snaith, 1983; German version: Herrmann-Lingen, Buss, & Snaith, 2005) | 18 months
  The measure assesses depression and anxiety.
Insomnia Severity Index (ISI; Bastien, Vallière, & Morin, 2001; German version: Pillmann, 2004) | 18 months
  The measure assesses the quality of sleep (sleep duration, sleep quality and negative impact on daily functioning).
Tinnitus Cognitions Questionnaire (T-Cog; Hiller & Haerkötter, 2005) | 18 months
  The measure assesses dysfunctional beliefs and cognitions regarding the tinnitus.
Tinnitus Acceptance Questionnaire (TAQ; Westin, Hayes, & Andersson, 2008; self-translated) | 18 months
  The measure assesses psychological acceptance of the tinnitus.
Anxiety Sensitivity Index - 3 (ASI-3; Taylor et al., 2007; German version: Kemper, Ziegler, & Taylor, 2007) | 18 months
  The measure assesses the fear of anxiety-related sensations.
Fear Avoidance Questionnaire (FAQ; self-developed measure) | 18 months
  The measure assesses fear-avoidance beliefs and behavior.
Working Alliance Inventory - Short Revised (WAI-SR; Horvath & Greenberg, 1986, 1989; German version: Wilmers et al., 2008) | 2 months
  The measure assesses three aspects of the therapeutic alliance (development of an affective bond, agreement on the tasks of therapy and agreement on the goals of therapy).
Credibility Scale (Devilly & Borkovec, 2000; self-translated and adapted to an intervention for tinnitus) | 6 months
  The scale assesses treatment credibility.
Therapy Expectancy Scale (self-developed) | baseline
  The scale assesses therapy expectancy.
Therapy Satisfaction Scale (self-developed) | week 10
  The scale assesses treatment satisfaction.
Web Screening Questionnaire for Common Mental Disorders (WSQ; Donker, van Straten, Marks, & Cuijpers, 2009; self-translated German version) | 3 months
  The questionnaire screens for depressive disorder, alcohol abuse/dependence, generalized anxiety disorder, posttraumatic stress disorder, social phobia, panic disorder, agoraphobia, specific phobia, and obsessive-compulsive disorder.
Big Five Inventory (BFI-10; Rammstedt & John, 2007; German version: Rammstedt & John, 2007) | baseline
  The measure is the short version of the Big Five Inventory (BFI; John, Donahue, & Kentle, 1991) and assesses the five personality traits extraversion, agreeableness, conscientiousness, neuroticism, and openness.
Process evaluation items (self-developed) | 18 months
  10 items assessing tinnitus loudness, tinnitus annoyance, perceived control, general mood, tinnitus acceptance, social functioning, behavioral avoidance and fear of sounds as well as the use of learned methods during the last week.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Hiller, Ph.D., Study Chair — Johannes Gutenberg University Mainz; Maria Kleinstäuber, Ph.D., Principal Investigator — Johannes Gutenberg University Mainz
Locations (1):
- Department of Clinical Psychology and Psychotherapy, Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Andersson G, Stromgren T, Strom L, Lyttkens L. Randomized controlled trial of internet-based cognitive behavior therapy for distress associated with tinnitus. Psychosom Med. 2002 Sep-Oct;64(5):810-6. doi: 10.1097/01.psy.0000031577.42041.f8. PMID 12271112
- [Background] Hiller W, Haerkotter C. Does sound stimulation have additive effects on cognitive-behavioral treatment of chronic tinnitus? Behav Res Ther. 2005 May;43(5):595-612. doi: 10.1016/j.brat.2004.03.012. PMID 15865915
- [Background] Kaldo V, Cars S, Rahnert M, Larsen HC, Andersson G. Use of a self-help book with weekly therapist contact to reduce tinnitus distress: a randomized controlled trial. J Psychosom Res. 2007 Aug;63(2):195-202. doi: 10.1016/j.jpsychores.2007.04.007. PMID 17662757
- [Background] Kaldo V, Levin S, Widarsson J, Buhrman M, Larsen HC, Andersson G. Internet versus group cognitive-behavioral treatment of distress associated with tinnitus: a randomized controlled trial. Behav Ther. 2008 Dec;39(4):348-59. doi: 10.1016/j.beth.2007.10.003. Epub 2008 Apr 20. PMID 19027431
- See also: Study registration website — http://www.kbt.info/mint/tinnitus.php